CLINICAL TRIAL: NCT06406738
Title: The Effect of High Reality Simulator Use in Newborn First Care Training on the Knowledge, Skills, Satisfaction and Self-Confidence of Midwifery Students
Brief Title: Simulator Use in Newborn First Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Sümeyye BAL, Director, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/3
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Newborn; Vitality
MeSH Terms: interventions — Models, Biological

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Reality Simulator (Experimental): Newborn first-care training will be given by the responsible investigator, and then one of the groups will be allocated by randomization. Using High Reality Simulator will perform Newborn first-care. These trainings will first be in the form of the instructor responsible for the groups demonstrating the application, and then the students will apply it one by one.
  Interventions: Other: Using High Reality Simulator
- control group (No Intervention): Using model will perform Newborn first-care. These trainings will first be in the form of the instructor responsible for the groups demonstrating the application, and then the students will apply it one by one.

INTERVENTIONS:
Other: Using High Reality Simulator — Using High Reality Simulator will perform newborn first-care.
  Other Names: model
  Arms: High Reality Simulator

SUMMARY:
The aim of this study is to determine the effects of using high-fidelity simulators in newborn first care training on the knowledge, skills, satisfaction and self-confidence of midwifery students.

DETAILED DESCRIPTION:
Hypotheses H01: There will no difference between the students' knowledge skills, satisfaction, and self-confidence of the simulation-based newborn first care training group and the knowledge skills, satisfaction, and self-confidence score of control group.

The study will be carried out in two different groups. The practice will start with meeting the students who apply to the study. After the students are evaluated in terms of eligibility criteria for the research, the students who are eligible will be informed about the research and written informed consent will be obtained from the women who accept. The random distribution of women to the study groups will be carried out using the Block Randomization method. The following applications will be made to the groups.

Newborn first care training will be given by the responsible investigator, and then one of the groups separated by randomization will perform newborn first care on the second group model using High Reality Simulator. These trainings will first be in the form of the instructor responsible for the groups demonstrating the application, and then the students will apply it one by one.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the research and obtaining written permission,

Exclusion Criteria:

-

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-06-29 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
First Care of the Newborn Information Form | immediately before simulation and immediately after the training and 6 weeks later
  t is a material developed by Karaçam Z, Çoban A, Taşpınar A (2018), consisting of 25 questions, to measure the student's knowledge level about newborn care. the minimum score is 0 and maximum score is 75.

CONTACTS AND LOCATIONS:
Overall Officials: Sumeyye BAL, Ph.D., Study Director — Ondokuz Mayıs University
Locations (1):
- Sumeyye, Ilkadim, Samsun, Turkey (Türkiye)